CLINICAL TRIAL: NCT03235583
Title: Validation of MotionPODTM a Device for Measuring Physical Activity, in Free-living Conditions
Brief Title: MOTIONPODTM Validation in Free-living Conditio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011.702
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-07

CONDITIONS: Obese; Healthy Volunteers
Keywords: Energy expenditure; physical activity; accelerometer; magnetometer; monitoring; free-living conditions; doubly labelled water
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MotionPod Validation (Other): Medical device validation
  Interventions: Device: MOTIONPODTM device validation

INTERVENTIONS:
Device: MOTIONPODTM device validation — MOTIONPODTM validation in free-living conditions using gold standards, including the DLW method

SUMMARY:
In this study, the investigators propose to assess the validity in measuring physical activity (PA) of a new PA monitor system the MOTIONPODTM, that coupled a hip-worn multi-sensor device (associating a tri-axial accelerometer, a magnetometer and a gyroscope) with an automatic activity/posture recognition algorithm and an activity-specific multilinear prediction model. The MOTIONPODTM performances in predicting mean daily PA energy expenditure (PAEE) will be calculated against the reference PAEE gold standard measure, using the doubly labeled water method (DLW). The MOTIONPODTM performances in predicting PAEE and PA patterns will be compared to those of two existing activity or movement monitors: the triaxial accelerometer ActigraphGT3X+TM and a device combining cardiofrequencemetry with accelerometry, the ActiheartTM. This latter has demonstrated fair performances but at the cost of a calibration of the heart-rate/EE relationship that limits its use in large population samples. Briefly, this open study will include 120 subjects, aged 18 to 75 years of both gender and with broad range of body mass index and physical activity level. The subjects will carry a MOTIONPODTM, an ActigraphGT3X+TM, an ActiheartTM and a GPS for a total of 14 days in everyday life conditions and complete a physical activity diary. In half of the subjects, PA will be evaluated on a period of 14 days, with standard PAEE measured by DLW. The other 60 subjects will be studied twice, one month apart, to test the reproducibility of the measures.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Age : 18 to 75 years
* Patients or healthy volunteers
* 40 obese subjects (BMI ≥ 30 kg/m2), 40 non-obese (BMI <30 kg/m2) and active (PA level evaluated by the RPAQ questionnaire) subjects, 40 non-obese and sedentary subjects
* Absence of cardiac rate disorders

Exclusion Criteria:

* Subjects with acute disorders: cardiovascular or neoplastic, severe infection during 3 previous months
* Subjects with a pathology restricting the walking distance (confinement, distance <200 meters)
* Subjects with implants (Pacemaker, cardiac implant or another active implant)
* Claustrophobic subjects (for subjects participating to "doubly labelled water" protocol)
* Drug use that could affect energy expenditure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2012-04-02 (Actual); Primary Completion 2013-10-11 (Actual); Study Completion 2013-10-11 (Actual)

PRIMARY OUTCOMES:
Daily physical activity energy expenditure (PAEE) MOTIONPODTM prediction | PAEE measurement will be measured over the 14-day study-period (Modality A) or the two 8-day periods (Modality B)
  MotionPodTM predictions will be calculated with the newly developed algorithms to evaluate the concordance between the physical activity energy expenditure (PAEE) estimated by the MOTIONPODTM and that of 2 physical activity monitors: the Actigraph GT3X+TM and the ActiheartTM. The estimation of PAEE by MotionPodTM will be compared with the measure of PAEE by DLW (gold standard measure, primary outcome 2/), with the measure of PAEE by Actiheart TM (primary outcome 3/), and with the measure of PAEE by ActigraphGT3X+ TM (primary outcome 4/).
Daily physical activity energy expenditure (PAEE) using DLW (gold standard measure) (modality A) | PAEE measurement will be measured over the 14-day study-period (Modality A)
  Daily Total Energy Expenditure (TEE) and PAEE standards will be measured with the DLW reference method. Briefly Resting metabolic Rate (RMR) will be measured via indirect calorimetry using a ventilated open-hood metabolic cart after a 12h-overnight fast. TEE will be determined using a 14-day multipoint DLW protocol. After providing a baseline urine sample, subjects will ingest a premixed dose of H218O (10% enriched) and 2H2O (99.85% enriched) DLW. Equilibration will be assessed in urine samples collected at 4h and 5h post dose. Subsequent urine samples will be collected every two days of the 14 days of the protocol. 2H2 and 18O isotopic enrichment will be analyzed in quadruplicate by pyrolysis on an elemental analyzer (Flash HT; ThermoFisher) interfaced with an IRMS (Delta V, ThermoFisher).
Daily physical activity energy expenditure (PAEE) Actiheart TM estimates (modalities A & B) | PAEE measurement will be measured over the 14-day study-period (Modality A) or the two 8-day periods (Modality B)
  ActiheartTM PAEE predictions will be calculated using the Actiheart software.
Daily physical activity energy expenditure (PAEE) ActigraphGT3X+ TM estimates (modalities A & B) | PAEE measurement will be measured over the 14-day study-period (Modality A) or the two 8-day periods (Modality B)
  ActigraphGT3X+TM PAEE predictions will be calculated using the ActigraphGT3X+ TM software.

SECONDARY OUTCOMES:
Identification and classification of activity/posture patterns by the MOTIONPODTM device (assessed by confusion matrices) | PAEE activity patterns will be evaluated over the 14-day study-period (Modality A) or over the two 8-day periods (Modality B)
  Different activities corresponding to the activity/recognition algorithm will be identified and quantified using the activity diary. The recognition rate of activity typologies (lying, sitting, inactive standing, active standing, walking, biking) by the MOTIONPODTM will be compared to data of the physical activity diary (measures (secondary measure outcome 2/). Confusion matrices will be used to compare the diary measures (secondary measure outcome 2/) with the MOTIONPODTM outputs.
Identification and classification of activities/postures patterns collected in the activity diary | PAEE activity patterns will be evaluated over the 14-day study-period (Modality A) or over the two 8-day periods (Modality B)
  Different activities corresponding to the activity/recognition algorithm will be identified and quantified using the activity diary.
(BMI < or > 30 kg/m2). | Baseline (at inclusion)
  to evaluate de concordance of MOTIONPODTM predictions with standard measure according to activity level, as previously described by subgroups

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche en Nutrition Humaine Rhône-Alpes - Centre hospitalier Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No